CLINICAL TRIAL: NCT04350515
Title: Effects of Social Exclusion in The Context of Chronic Embitterment: How Social Exclusion Experiences Affect Chronic Embittered People in Their Behaviour and Physiology
Brief Title: Effects of Social Exclusion in The Context of Chronic Embitterment
Acronym: EMBEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: EMBEX
Record Dates: First submitted 2019-12-20; First posted 2020-04-17 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Emotional Stress; Embitterment
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyberball: Other Exclusion (Experimental): Cyberball Paradigm - the avatar will be excluded by the player
  Interventions: Other: Cyberball: Other Exclusion; Other: Mindfulness: Emotion Regulation Task; Other: Mindfulness: Word Recognition Task
- Cyberball: Player Exclusion (Experimental): Cyberball Paradigm - the player will be excluded by the other players
  Interventions: Other: Cyberball: Player Exclusion; Other: Mindfulness: Emotion Regulation Task; Other: Mindfulness: Word Recognition Task

INTERVENTIONS:
Other: Cyberball: Other Exclusion — A cyberball paradigm, whereas 2 avatars and the subject are playing a virtual ball tossing game. In this condition, one of the avatars is excluded.
  Other Names: In terms of outcome measure 'points for fairness': intervention condition; In terms of outcome measure 'changes in HRV': control condition
  Arms: Cyberball: Other Exclusion
Other: Cyberball: Player Exclusion — A cyberball paradigm, whereas 2 avatars and the subject are playing a virtual ball tossing game. In this condition, the subject is excluded by the avatars.
  Other Names: In terms of outcome measure 'points for fairness': control condition; In terms of outcome measure 'changes in HRV': intervention condition
  Arms: Cyberball: Player Exclusion
Other: Mindfulness: Emotion Regulation Task — In this task, subjects listen to an audio file containing a scripted emotion regulation exercise. This exercise is based by the authors Nissen & Sturm (2018). It takes around 14 minutes to complete the whole task.
  Other Names: Intervention Condition
Other: Mindfulness: Word Recognition Task — In this task, subjects listen to an audio file containing a scripted word recognition exercise. It contains both contrary words recognition (e.g. "The opposite of loud is ...") and completion of german sayings (e.g. "That's where the dog is..."). It takes around 14 minutes to complete the whole task.
  Other Names: Control Condition

SUMMARY:
This experimental, anonymous labor study aims to examine how experiences of social exclusion influence individuals in their fairness-behaviour, psychophysical reactions, and emotion regulation depending on their extent of bitterness. Points given for fairness reasons, just world belief, rejection sensitivity, well-being, cognitive emotion regulation strategies, and heart rate variability (HRV) are measured and analyzed using structural equation modeling and multiple regression.

DETAILED DESCRIPTION:
Embitterment is defined as an emotional response due to an event which is subjectively perceived as unjust. Nonetheless, there is little empiric evidence of unjust behaviour by others in the interpersonal context that triggers embitterment reactions. Ostracism, is an act where a person is excluded from a social environment without any reasons. This experimental labor study examines how the experiences of this form of social exclusion influences individuals depending on their self-evaluated embitterment. That is, fairness-behaviour is assessed as well as changes in hearth rate variability.

ELIGIBILITY:
Inclusion Criteria:

* German language, 18 years old, no cardiovascular disease
* The participation in the anonymous labor study is voluntary, participants gave consent to use the data with their participation.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Points for Fairness | After the second Cyberball intervention (exclusion of the subject or the avatar), at approx. 30 minutes from baseline.
  Asked after the second Cyberball game session. Each participant will be asked, how many of their "earned" points (from the first Cyberball round) they are willing to compensate for fairness reasons towards the group. This is assessed by a Likert scale ranging from 0 - 14; giving zero points it the least one can give, 14 is the maximum.
Changes in Heart Rate Variability (HRV; RMSSD) from baseline (t0) | After approx. 15, 20, 25, 30, 35, 40, 45, and 50 minutes from baseline.
  Changes in Heart Rate Variability (RMSSDs) are assessed using the hardware of BIOPAC Systems. The extraction and analysis of the RMSSDs are performed with Kubios HRV premium (software).

SECONDARY OUTCOMES:
Belief in a Just World | Baseline questionnaires at the beginning of the experiment.
  Belief in a Just World is assessed using the german version of the "Beliefs in a just world questionnaire" (Dalbert, Montada, & Schmitt, 1987). It contains six items, ranging from 1-6, whereas lower numbers indicate a lower belief in a just/rightful world and vice versa.
Rejection Sensitivity | Baseline questionnaires at the beginning of the experiment.
  Rejection Sensitivity is assessed using the german version of the "Rejection Sensitivity Questionnaire" (Feldman & Downey, 1994) - based on 18 items describe interpersonal interactions, where the subject has to ask someone to do something for him or her, further how much distress these interactions would provoke and the other person would decline the request. Each item can be answered on a Likert-Scale from 1-6, whereas lower numbers indicate less personal distress and expected rejection by the interacting person when being in that particular scenario. Higher Numbers indicate more distress from the scenario as well as the more is a rejection expected.
Cognitive Emotion Regulation (Strategies) - Basic | Baseline questionnaires at the beginning of the experiment.
  Emotion Regulation are assessed using the german version of the "Emotion Regulation Questionnaire" (ERQ; Gross & John, 2003; Abler & Kessler, 2011). This questionnaire assesses basic tendencies of the two strategies "reappraisal" and/or "Suppression" with regards to emotion regulation. It has 10 items which can be answered based on a Likert-Scale ranging from 1 - 7. The higher the number the more the person tends to use this particular strategy and vice versa.
Cognitive Emotion Regulation (Strategies) - Specific | Baseline questionnaires at the beginning of the experiment.
  Specific Cognitive Emotion Regulation Strategies are assessed using the german version of the Cognitive Emotion Regulation Questionnaire (CERQ; Garnefski, Kraaij & Spinhoven, 2001). This questionnaire assesses nine dimensions of cognitive coping styles (e.g. "other-blame") in response to distress. It contains 36 items which can be answered on a Likert-Scale ranging from "(almost) never" (0) to "(almost) every time" (4). Higher number indicate the higher the tendency of usage of the specific strategy and vice versa.
Mindfulness Experiences | Baseline questionnaires at the beginning of the experiment.
  Mindfulness Experiences is assessed using the Comprehensive Mindfulness Scale (CHIME; Bergomi, Tschacher, & Kupper, 2014). It assesses different aspects of mindfulness experiences in daily life based on 37 items, ranging from 0 - 5. Higher number indicate the higher the awareness towards the particular experience and vice versa.
Change from baseline in subject's well-being - overall | After 15, 20, 30, 45, and 50 minutes from baseline.
  Overall subjective well-being is assessed by asking the participant five times "How do you feel right now?" The subject can answer by the use of a bipolar scale (-2 "very bad", 0 "neutral", +2 "very good").
Change from baseline in subject's well-being - specific | After the mindfulness task (50 minutes) from baseline
  Specific subjective well-being is assessed the "Mehrdimensionale Befindlichkeitsfragebogen" (MDBF; Steyer, Notz, Schwenkmezger, & Michael Eid, 1997). This questionnaire contains 24 items and measures on three bipolar dimensions (mood, vigilance, and distress) present mental state. Answers can be made on a Likert-Scale ranging from "absolutely not" (-2) till "very much" (+2). The lower the number the worse the mood, or the weariness, or the distress, depending on the dimension, and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Koroma, M.Sc., Principal Investigator — University of Bern, Department of Psychology
Locations (1):
- University of Bern, Institute of Psychology, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://embex.unibe.ch